CLINICAL TRIAL: NCT05499442
Title: Construction of Non-invasive EEG Motor Movement and Imagery Dataset for Stroke
Brief Title: EEG Motor Movement and Imagery Dataset for Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: haojunwei8
Record Dates: First submitted 2022-04-01; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators collect and analyze the alpha and beta wave of EEG activity at the motor cortices of the participants, When the motor task is being performed. The Brodmann area 10-20 method and portable EEG equipment was used in the single-center study.

DETAILED DESCRIPTION:
To understand the motor mechanism of stroke patients with motor dysfunction, an EEG motor movement and imagery dataset for Stroke will be created. 120 subjects will be enrolled in the single-center study. The investigators collect and analyze the EEG activity at the motor cortices of the participants, When the motor movement or imagery task is being performed. The alpha and beta wave of EEGs were recorded from 32 electrodes as per the international 10-20 system with portable EEG equipment.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of cerebral infarction conforms to the diagnostic criteria of Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2018, and the diagnosis of intracerebral hemorrhage conforms to the diagnostic criteria of Chinese guidelines for the diagnosis and treatment of intracerebral hemorrhage 2019.
2. First onset.
3. Age ≥ 18 years old.
4. Motor dysfunction of upper and / or lower limbs: muscle strength decreased by 0 to 5-grade and / or ataxia.
5. Informed consent has been signed.

Exclusion Criteria:

1. Vital signs are unstable.
2. Serious circulatory system, respiratory system, motor system and other diseases, such as atrial fibrillation, heart failure, pulmonary infection, severe liver and kidney insufficiency, lower extremity venous thrombosis and other serious diseases.
3. Functional impairment of upper or lower limbs caused by other diseases of nervous system or other reasons, such as fracture, deformity, etc.
4. Unable to cooperate to complete the examination, such as mental disorder, cognitive impairment, visual impairment, sitting balance disorder, etc
5. Other reasons: alcoholism; Skull defect; Head skin defect, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with motor dyfunction in Xuanwu Hospital of Capital Medical University were admitted from January 1, 2022 to December 31, 2023
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG characteristics of motor | 1-7day
  EEG Characteristics for Motor Execution and Motor Imagery
Action Research Arm Test | 1-7days
  Use the assessment scale of Action Research Arm Test evaluation completes the limb function evaluation
Fugl-meyer Assessment | 1-7days
  Use the assessment scale of Fuel-meyer to evaluate completes the limb function evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing, Beijing Municipality, China